CLINICAL TRIAL: NCT04080856
Title: Real-World Experience of Elagolix For the Treatment of Endometriosis in Canada: An Observational Cohort Study (GRACE)
Brief Title: Real-World Experience Study of Elagolix For the Treatment of Endometriosis in Canada
Acronym: GRACE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P19-933
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Endometriosis
Keywords: Endometriosis; Elagolix; Real-World; Effectiveness
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with endometriosis: Premenopausal participants with endometriosis receiving elagolix in real-world setting

SUMMARY:
The objective of this study is to evaluate real-world effectiveness of elagolix in Canadian women with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed elagolix as part of standard treatment
* Naive to elagolix prior to starting this study or have stopped taking elagolix for 2 months prior to the start of this study
* Symptomatic endometriosis (clinically or surgically diagnosed) including currently experiencing dysmenorrhea
* Has provided written informed consent allowing the use of their data for the study

Exclusion Criteria:

* Did not consent
* Cannot fill out questionnaires
* Prescribed elagolix for a period of 1 or 2 months only
* Post-menopausal (naturally or surgically)
* Symptomatic uterine fibroid(s)
* Had medical treatment for uterine fibroids (any length of treatment)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Premenopausal participants with endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Change in Dysmenorrhea Score | From Baseline (Month 0) to Month 6
  Dysmenorrhea is evaluated through 11-point numeric rating scale (NRS), where 0 = no pain and 10 = worst imaginable pain

SECONDARY OUTCOMES:
Percentage of Participants With Patient Global Impression of Change (PGIC) Response | Up to approximately 18 months
  PGIC is a questionnaire-based assessment of endometriosis-related pain is since initiation of study drug.
Percentage of Participants With Clinician's Global Impression of Change (CGIC) Response | Up to approximately 18 months
  CGIC score is summarized assessment of clinical diagnosis of patient's illness by clinician in relative to a baseline state.
Change From Baseline in Non-Menstrual Pelvic Pain (NMPP) | From Baseline (Week 0) to approximately 18 months
  The NMPP pain scale ranges from 0 (none) to 3 (severe) as recorded in a daily electronic diary.
Change From Baseline in Dyspareunia Score | From Baseline (Week 0) to approximately 18 months
  Dyspareunia pain scale ranges from 0 (absent) to 3 (severe).
Change From Baseline in Pelvic Pain During Periods | From Baseline (Week 0) to approximately 18 months
  Change in pelvic pain is patient reported questionnaire to rate the severity of pelvic pain during periods on the scale of 0 to 10, where 0 = no pain and 10 = worst imaginable pain.
Change from Baseline in Bleeding and Menstrual Cycle | From Baseline (Week 0) to approximately 18 months
  Uterine bleeding was reported by participants during the study using the e-Diary.
Percentage of Participants With Change in Dosing Schedule | Up to approximately 18 months
  Percentage of participants who change dose as well as the reasons for change will be tabulated.
Change from Baseline in Morisky Medication Adherence Scale (MMAS) | From Baseline (Week 0) to approximately 18 months
  The Morisky Medication Adherence Scale (MMAS) is a 4-item questionnaire assessing the risk of non-adherence to medications.
Percentage of Participants Using Concomitant Medications/Treatments | Up to approximately 18 months
  Percentage of participants using concomitant medications/treatments is assessed.
Percentage of Participants Using Other Medications/Treatments | Up to approximately 18 months
  Percentage of participants using other medications/treatments for endometriosis is assessed.
Percentage of Participants Using Pain/Rescue Medications | Up to approximately 18 months
  Percentage of participants using pain/rescue medications is assessed.
Percentage of Participants Using Add-Back | Up to approximately 18 months
  Percentage of participants with use of add-back is reported
Change from Baseline in Endometrial Health Profile (EHP)-30 | From Baseline (Week 0) to approximately 12 months
  EHP-30 is a disease-specific self-administered questionnaire used to measure health related QoL in women with endometriosis. EHP-30 covers 5 dimensions: pain, control and powerlessness, social support, emotional wellbeing, and self-image.
Change from Baseline in Endometrial Health Profile (EHP)-5 | Up to approximately 6 months post-treatment (Month 12)
  EHP-5 is a disease-specific self-administered questionnaire used to measure health related QoL in women with endometriosis.
Change from Baseline in Work Productivity and Activity Impairment (WPAI) | From Baseline (Week 0) to approximately 18 months
  WPAI questionnaire is used to measure the effect of general health and symptom severity on work productivity and regular activities during the past seven days.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (18):
- Canada (18):
  - South Health Campus Rheumatology Clinic /ID# 213065, Calgary, Alberta
  - Aubrey D. Uretsky Professional Corporation /ID# 214753, Edmonton, Alberta
  - BC Women's Hospital /ID# 214561, Vancouver, British Columbia
  - Strand Clinic /ID# 213567, St. John's, Newfoundland and Labrador
  - IWK Health Center /ID# 213066, Halifax, Nova Scotia
  - Medicor Research Inc /ID# 213467, Greater Sudbury, Ontario
  - Hamilton Health Sciences - McMaster University Medical Centre /ID# 213496, Hamilton, Ontario
  - Dr. George A. Vilos Medicine Professional Corporation /ID# 214497, London, Ontario
  - Ottawa Hospital Research Institute /ID# 213608, Ottawa, Ontario
  - Sunnybrook Health Sciences Ctr /ID# 214330, Toronto, Ontario
  - Unity Health Toronto - St. Michael's Hospital /ID# 213590, Toronto, Ontario
  - CISSS - Hôpital de Gatineau /ID# 212944, Gatineau, Quebec
  - Jessima R&D Inc. /ID# 212943, LaSalle, Quebec
  - Clinique de Gynecologie-Obstetrique Pierre Boucher /ID# 213064, Longueuil, Quebec
  - CIUSSS de l'est de l'Ile-de-Montreal - Hopital Maisonneuve-Rosemont /ID# 213439, Montreal, Quebec
  - Jewish General Hospital /ID# 215728, Montreal, Quebec
  - Duplicate_Brunswick Medical /ID# 214743, Montreal, Quebec
  - CHU de Quebec-Université Laval hôpital CHUL /ID# 213677, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P19-933&Latitude=&Longitude=&LocationName=#additional-resources-section